CLINICAL TRIAL: NCT07268040
Title: A Multicenter, Open-label Phase II Clinical Study of SHR-7787 Combined With Other Antitumor Drugs in Patients With Advanced Solid Tumors
Brief Title: A Trial of SHR-7787 Injection Combined With Other Anti-tumor Drugs in Patients With Malignant Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-7787-201
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Tumors
MeSH Terms: interventions — Etoposide; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SHR-7787 combined with SHR-1316 (Experimental): SHR-7787 injection combined with SHR-1316 injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-1316 Injection
- SHR-7787 combined with SHR-4849 (Experimental): SHR-7787 injection combined with SHR-4849 injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-4849 Injection
- SHR-7787 combined with etoposide and carboplatin/cisplatin (Experimental): SHR-7787 injection combined with etoposide and carboplatin/cisplatin injection.
  Interventions: Drug: SHR-7787 Injection; Drug: Etoposide injection; Drug: Carboplatin injection; Drug: Cisplatin injection
- SHR-7787 combined with SHR-1316, etoposide, carboplatin/cisplatin (Experimental): SHR-7787 injection combined with SHR-1316, etoposide, carboplatin/cisplatin injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-1316 Injection; Drug: Etoposide injection; Drug: Carboplatin injection; Drug: Cisplatin injection
- SHR-7787 combined with SHR-4849 and SHR-1316 (Experimental): SHR-7787 injection combined with SHR-4849 and SHR-1316 injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-1316 Injection; Drug: SHR-4849 Injection
- SHR-7787 combined with SHR-1316 and BP102 (Experimental): SHR-7787 injection combined with SHR-1316 and BP102 injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-1316 Injection; Drug: BP102 Injection
- SHR-7787 combined with SHR-4849 and BP102 (Experimental): SHR-7787 injection combined with SHR-4849 and BP102 injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-4849 Injection; Drug: BP102 Injection
- SHR-7787 combined with SHR-4849, SHR-1316 and carboplatin/cisplatin (Experimental): SHR-7787 injection combined with SHR-4849, SHR-1316 and carboplatin/cisplatin injection.
  Interventions: Drug: SHR-7787 Injection; Drug: SHR-1316 Injection; Drug: SHR-4849 Injection; Drug: Carboplatin injection; Drug: Cisplatin injection

INTERVENTIONS:
Drug: SHR-7787 Injection — SHR-7787 Injection.
Drug: SHR-1316 Injection — SHR-1316 Injection.
  Arms: SHR-7787 combined with SHR-1316; SHR-7787 combined with SHR-1316 and BP102; SHR-7787 combined with SHR-1316, etoposide, carboplatin/cisplatin; SHR-7787 combined with SHR-4849 and SHR-1316; SHR-7787 combined with SHR-4849, SHR-1316 and carboplatin/cisplatin
Drug: SHR-4849 Injection — SHR-4849 Injection.
  Arms: SHR-7787 combined with SHR-4849; SHR-7787 combined with SHR-4849 and BP102; SHR-7787 combined with SHR-4849 and SHR-1316; SHR-7787 combined with SHR-4849, SHR-1316 and carboplatin/cisplatin
Drug: Etoposide injection — Etoposide Injection.
  Arms: SHR-7787 combined with SHR-1316, etoposide, carboplatin/cisplatin; SHR-7787 combined with etoposide and carboplatin/cisplatin
Drug: Carboplatin injection — Carboplatin Injection.
  Arms: SHR-7787 combined with SHR-1316, etoposide, carboplatin/cisplatin; SHR-7787 combined with SHR-4849, SHR-1316 and carboplatin/cisplatin; SHR-7787 combined with etoposide and carboplatin/cisplatin
Drug: Cisplatin injection — Cisplatin Injection.
  Arms: SHR-7787 combined with SHR-1316, etoposide, carboplatin/cisplatin; SHR-7787 combined with SHR-4849, SHR-1316 and carboplatin/cisplatin; SHR-7787 combined with etoposide and carboplatin/cisplatin
Drug: BP102 Injection — BP102 Injection.
  Arms: SHR-7787 combined with SHR-1316 and BP102; SHR-7787 combined with SHR-4849 and BP102

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of SHR-7787 in combination with other anti-tumor drugs in patients with malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study;
2. Patients with histologically or cytologically confirmed unresectable solid tumors;
3. At least one measurable lesion was identified per RECIST 1.1;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
5. Adequate organ functions as defined per protocol;
6. Minimum life expectancy of 3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) metastases;
2. History of other malignancy within the past 5 years, with exceptions defined in the protocol;
3. Patients with uncontrolled cancer pain;
4. Patients with serious cardiovascular and/or cerebrovascular diseases;
5. Uncontrollable third-space effusion, such as pleural effusion, pericardial effusion or peritoneal effusion;
6. Patients with Severe infections within 4 weeks prior to the first dose;
7. Active pulmonary tuberculosis infection;
8. History of immunodeficiency;
9. History of autoimmune diseases;
10. The adverse events of previous antineoplastic therapy did not recover to CTCAE≤ grade 1;
11. Pregnant or nursing women, or planned to become pregnant during the study period;
12. Known allergic to any component of investigational drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The Recommended phase II dose of SHR-7787 injection monotherapy (stage I) | Expected to be two years after the start of the study.
Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (stage I) | About 1 year after study initiation.
Incidence and severity of serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (stage I) | About 1 year after study initiation.
Incidence of Dose Limited Toxicity (DLT) described in the protocol (stage I) | About 1 year after study initiation.
Objective response rate (ORR) (stage II) | Expected to be two years after the start of the study.
Progress Free Survival (FPS) (stage II) | Expected to be two years after the start of the study.

SECONDARY OUTCOMES:
Objective response rate (ORR) | About 1 year.
Duration of Response (DoR) | About 1 year.
Disease Control Rate (DCR) | About 1 year.
Progress Free Survival (PFS) | About 1 year.
Overall Survival (OS) | About 1 year.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided